CLINICAL TRIAL: NCT05748457
Title: Changes in Outcomes of Treatment for Adolescent Anorexia Nervosa After Implementation of Family Based Treatment in a Norwegian Child and Adolescent Mental Health Service: A Retrospective Cohort Study With Prospective Follow-up
Brief Title: Akershus University Hospital Retrospective Cohort Study of Family Based Treatment
Acronym: ARCS-FBT
Status: Terminated | Type: Observational
Why Stopped: The proportion of eligible participants consenting was too low (21%) too draw any conclusions.
Sponsor: University Hospital, Akershus (Other)
Collaborators: Rådgivning om Spiseforstyrrelser (Unknown)
Responsible Party: Principal Investigator, Erling W. Rognli, Psykologspesialist, University Hospital, Akershus
Other Study IDs: 2021_182
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2015-2017: Patients treated for anorexia nervosa in the years 2015-2017 at Nedre Romerike outpatient clinic, Department of child and adolescent mental health services, Akershus university hospital.
  Interventions: Behavioral: Non-manualised family therapy.
- 2018-2020: Patients treated for anorexia nervosa in the years 2018-2020 at Nedre Romerike outpatient clinic, Department of child and adolescent mental health services, Akershus university hospital.
  Interventions: Behavioral: Family Based Treatment

INTERVENTIONS:
Behavioral: Non-manualised family therapy. — Family therapy provided by qualified therapists without reference to a specific therapy manual.
  Groups: 2015-2017
Behavioral: Family Based Treatment — Family therapy implemented according to the published "Treatment manual for anorexia nervosa: A family-based approach" by Lock & Le Grange (2nd edition, 2015).
  Groups: 2018-2020

SUMMARY:
The goal of this observational study is to compare short and long-term effects of manualised Family Based Treatment for adolescent anorexia nervosa to those of non-manualised family therapy. The study will approach former patients who were treated before and after Family Based Therapy was adopted in an outpatient clinic, and extract data from electronic health records and public registries.

DETAILED DESCRIPTION:
A two-group retrospective exploratory cohort study with longitudinal follow-up comparing adolescents with anorexia nervosa treated with generic family therapy to those treated with the manualised Family Based Treatment (FBT). The primary aim is to investigate whether adoption of FBT has led to faster normalisation of weight and lower rates of eating disorder in early adulthood. Secondary aims are to investigate whether implementation of FBT has changed the time to discharge, heterogeneity of patient weight change across treatment, rates of adverse events, rates of readmission, patient experiences of the treatment, long term functional outcomes and mortality. Data are extracted from patient health records, reported by participants and extracted from public registries.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of F50.0 Anorexia nervosa or F50.1 Atypical anorexia nervosa according to the International Classification of Diseases-10.

Exclusion Criteria:

• Patient was treated during the years 2018-2020 and FBT was never initiated according to patient health records.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients initiating treatment during the years 2015-2020 with the eating disorder team at Nedre Romerike outpatient clinic at Akershus university hospital, Department of child and adolescent mental health services.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Time to weight restoration | Assessed retrospectively at enrolment.
  Number of days from start of treatment to a weight measurement placing the patient at or above 95% of expected body weight (50. percentile) for age and sex given Norwegian population norms.

SECONDARY OUTCOMES:
Time to discharge from treatment | Assessed retrospectively at enrolment.
  Number of days from start of treatment to the date of discharge from the outpatient clinic.
Time to readmission to treatment | Assessed retrospectively at enrolment.
  Number of days from start of treatment to any date of readmission to the outpatient clinic.
Mortality | Assessed 5, 10, 15 and 20 years post treatment.
  Death from any cause.
Level of education | Assessed 5, 10, 15 and 20 years post treatment.
  Highest level of education achieved, obtained from national registries.
Employment status and welfare benefits | Assessed 5, 10, 15 and 20 years post treatment.
  Employment status or receipt of welfare benefits, obtained from national registries.
Treatment for eating disorder in adulthood | Assessed 5, 10, 15 and 20 years post treatment.
  Treatment in specialist mental health services for any eating disorder.

OTHER OUTCOMES:
Participant experiences and satisfaction with services | Assessed retrospectively at enrolment.
  Generic Short Patient Experiences Questionnaire (GS-PEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Erling W Rognli, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Nedre Romerike BUP, Lillestrøm, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared for legal reasons.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT05748457/Prot_SAP_000.pdf